CLINICAL TRIAL: NCT04279587
Title: Camp Based Multi-component Intervention for Families of Young Children With Type 1 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to COVID-19 pandemic
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Olga Gupta, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0282
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Residential camp participant (Experimental): Participants will attend a 3 day family-centered, multidisciplinary, intensive education session at a regional camp.
  Interventions: Behavioral: Residential camp

INTERVENTIONS:
Behavioral: Residential camp — Intensive education at a residential camp.

SUMMARY:
Eighteen preschool aged children and their families will attend structured, multidisciplinary, family-centered intensive education sessions over a 3-day weekend in a residential camp setting to address the unique challenges of managing type 1 diabetes mellitus in young children.

DETAILED DESCRIPTION:
The invesigators propose to deliver a structured multidisciplinary family-centered intervention over a 3-day weekend. The intervention will be based at a regional camp. The proposed camp encounters aim to provide:

* An opportunity for intensive education beyond that achievable in a single class, and without the unfavorable impacts of multiple weekday classes on family and work time.
* Varied educational modalities including didactic sessions, practical demonstrations and role playing.
* Close observation of each child throughout the day and night by experienced diabetes counselors and medical staff to identify and help correct maladaptive family behaviors.
* A safe environment where parents can participate in group therapy sessions without child care worries.
* An opportunity for age-appropriate child-centered educational and therapeutic activities.
* An opportunity for families to form mutually-supportive friendships.
* Fun weekends away where the parents have help caring for their diabetic children.

The investigators will conduct this pilot study, which will enroll 18 preschool children age 3-5.5 years, with the goal of obtaining preliminary results for 15 subjects.

The primary outcome, to be determined approximately one month before and 3 months after the camp session, is improvement in Hemoglobin A1c (HbA1c).

Exploratory Hypotheses:

Compared with pretreatment baseline, subjects attending a 3-day session at a family diabetes camp will improve:

* HbA1c 3 months after the first camp session
* Behavioral/QoL assessments, including the parents of young children version of the hypoglycemia fear survey (HFS-P-YC), the Behavioral Pediatrics Feeding Assessment Scale (BPFAS), and the general and diabetes modules of the PedsQL.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-5.5 years old (+/- 2 months) at the date of camp session they are eligible to join.
* Child and Parents fluent in English
* Type 1 diabetes mellitus diagnosed for at least 10 months previous to date of first camp they are eligible to join.
* Taking insulin
* Custodial parent or guardian (preferable both parents or guardians) willing to attend both session of camp and the activities scheduled for them.
* Parent or guardian must sign consent before any study procedures are performed.

Exclusion Criteria:

* Neonatal diabetes (diagnosis in the first 3 months of life) or documented Monogenic Diabetes of Youth; i.e., a likely genetic form of diabetes rather than an autoimmune etiology.
* Post-surgical diabetes (e.g., pancreatectomy for congenital hyperinsulinism). Such patients often cannot secrete glucagon, leading to a particularly severe inability to defend against hypoglycemia.
* Other severe chronic disease (e.g., cancer, cystic fibrosis) which in the judgment of the investigator is likely to significantly affect glycemic control.
* Patients cannot be taking systemic corticosteroids at enrollment because of adverse effects on glycemic control, but the investigators will not disqualify subjects who require such therapy during the study. Inhaled or topical corticosteroids are permissible.
* Patients with hypothyroidism or hyperthyroidism must be clinically euthyroid and have free T4 and thyroid stimulating hormone within age-appropriate reference ranges at last medically indicated testing. Patients with out of range values may be retested after medication dose adjustment.
* Developmental delay or behavioral disorder in the patient of sufficient severity, in the judgment of the investigator, to interfere with group activities.
* Medical or psychiatric disorder in a parent of sufficient severity, in the judgment of the investigator, to interfere with group activities.
* Celiac disease is not an exclusion criterion.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | 3 months
  3 month marker of glycemic control

SECONDARY OUTCOMES:
Change in PedsQL Family Impact Module | 3 months
  Survey measure of impact the child's chronic disease has on the family
Change in PedsQL Pediatric Quality of Life Inventory | 3 months
  Survey measure of quality of life
Change in Hypoglycemia Fear Survey | 3 months
  Survey measure of hypoglycemia fear
Change in Behavioral Pediatrics Feeding Assessment | 3 months
  Survey measure of child feeding habits

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Perrin C White, Dallas, Texas
  - Children's Medical Center, Dallas, Texas